CLINICAL TRIAL: NCT03176121
Title: A Long Term, Open-Label, Multi-Center Study Evaluating Safety and Tolerability of Oxycodone in Patients With Moderate to Severe Cancer Pain
Brief Title: Study Evaluating Safety and Tolerability of Oxycodone in Patients With Moderate to Severe Cancer Pain
Acronym: STOP Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taiwan Mundipharma Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OXY16-TW-401
Record Dates: First submitted 2017-05-22; First posted 2017-06-05 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2017-06

CONDITIONS: Cancer; Pain
Keywords: Oxycodone; Cancer Pain; Long-term use
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oxycodone treatment (Experimental): Patients will take either control-released oxycodone (OxyContin® 10mg and 20mg) or immediate-released oxycodone (OxyNorm® 5mg) or both for initial dose and used it to titrate his/her background dose.
  After regular time assessment of the pain score (NRS), if the pain control is inadequate (NRS ≥ 4), a total daily dose in 24hrs will be summed up for the next dose titration until reach a stable dose (as defined as total daily dose is fixed for at least two weeks).
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — Patients will take either CR oxycodone or IR oxycodone or both for initial dose and used it to titrate his/her background dose.

SUMMARY:
This study is to evaluate the safety and tolerability of oxycodone control-released (CR) and/or immediate-released (IR) use in patients with moderate to severe cancer pain in a 3-months period in Taiwan.

DETAILED DESCRIPTION:
This is an open label, long-term study carrying in multi-centers. Around 200 patients with moderate to severe cancer pain (NRS ≥ 4) who agreed and signed informed consent will be enrolled to receive oxycodone with continuous around-the-clock pattern. The study is to evaluate the safety and tolerability of cancer patients who receive CR and/or IR oxycodone. The number and percentage of patients with adverse events and serious adverse events will be recorded throughout the study.

The study will continue for 3 months to observe the safety and tolerability. After screening at Screening visit, patients begin the study by the first day visit (Day 1). Pain assessment, study related questionnaires are giving out to measure the baseline scale of each patient. Questionnaires including rate of quality of analgesia, EQ-5D and clinical opiate withdrawal scale (COWS). The prescription of the study drug will be recorded from Day 1. Patients will need to visit bi-weekly, including Wk 2 (Day 14±3), Wk 4 (Day 28±3), Wk 6 (Day 42±3), Wk 8 (Day 56±3), Wk 10 (Day 70±3) and Wk 12 (Day 84±3). Pain assessment will be assessed in each visit, drug accountability will be recorded accordingly. The rate of quality of Analgesia will be assessed in each visit; QoL (EQ-5D) will be recorded in Wk 4, Wk 8 and Wk 12. The COWS will be assessed again in Wk 12.

The safety for individual patient will be followed during study up to 2 weeks after the end of treatment (EOT) or early termination (ET). The telephone contact for safety follow-up is acceptable for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients aged 20 years old and over
2. ECOG ≤ 2
3. Moderate to severe pain intensity (NRS pain score ≥ 4)
4. Cancer-related pain that requires treatment with continuous around-the-clock strong opioid analgesic
5. Patients who will not be treated with radiotherapy within 7 days prior to screening and during study
6. Patients or his/her caregivers who are able to fill out the questionnaire forms
7. Patient provided signed informed consent

Exclusion Criteria:

1. Patients diagnosed with non-cancer pain or unexplained pain
2. Patients who cannot be applicable for oral administration
3. Patients who have constipation (CTCAE grade 3 and above)
4. Patients with evidence of significant structural/functional abnormalities of GI tract or planned to undergo surgeries that have high risk lead to gastrointestinal stenosis, blind loop or gastrointestinal obstruction during study
5. Abnormal lab results, with obvious clinical significance, such as the creatinine ≥ 2 fold of upper limit of normal value, or ALT or AST ≥ 2.5 fold of upper limit of normal value (≥ 5 fold, to the patients with liver metastasis or primary liver cancer), or liver function of Child C grade prior to study
6. Pregnant or nursing (lactating) women
7. Patients who are drug or alcohol abuse
8. Patients with moderate to severe psychiatric problems
9. Patients who have hypersensitivity to oxycodone
10. Patients who are clinically unstable or have a life expectancy of less than three months making completion of the trial unlikely

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number and percentage of patients with adverse events (AEs) and serious adverse events (SAEs) | Up to 14 weeks
  Number and percentage of patients with adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Change from baseline pain intensity scale (NRS) | Up to 12 weeks
  The change from baseline pain intensity scale (NRS) to each visit
Time (days) needs in first titration to a stable dose | Up to 12 weeks
  The time (days) needs in first stable titration
Average dosage (mg/day) needs in first titration to a stable dose | Up to 12 weeks
  The average dosage needs in first stable titration
Quality of analgesia using rating of excellent, very good, good, fair or poor | Up to 12 weeks
  The percentage of patients rating quality of analgesia of excellent, very good, good, fair or poor
Treatment discontinuation reason (due to AE, withdraw consent, or any kinds of reasons) | Up to 12 weeks
  Analysis treatment discontinue reason (due to AE, withdraw consent, or any kinds of reasons)
Change from baseline in QoL questionnaire (EQ-5D) | Up to 12 weeks
  The change from baseline in QoL questionnaire (EQ-5D)
Opiate withdrawal level by Clinical Opiate Withdrawal Scale (COWS) | Up to 12 weeks
  The change of clinical opiate withdrawal scale (COWS) from baseline
Safety and tolerability (PE and vital sign change from baseline) | Up to 14 weeks
  The change from baseline in PE and vital sign

CONTACTS AND LOCATIONS:
Locations (10):
- Taiwan (10):
  - Changhua Christian Hospital, Chang-hua
  - Chang Gung Memorial Hospital, Chiayi branch, Chiayi City
  - Chang Gung Memorial Hospital, Kaohsiung branch, Kaohsiung City
  - Chang Gung Memorial Hospital, Keelung branch, Keelung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - MacKay Memorial Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, LinKou branch, Taoyuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Breivik H, Cherny N, Collett B, de Conno F, Filbet M, Foubert AJ, Cohen R, Dow L. Cancer-related pain: a pan-European survey of prevalence, treatment, and patient attitudes. Ann Oncol. 2009 Aug;20(8):1420-33. doi: 10.1093/annonc/mdp001. Epub 2009 Feb 24. PMID 19244085
- [Background] Caraceni A, Hanks G, Kaasa S, Bennett MI, Brunelli C, Cherny N, Dale O, De Conno F, Fallon M, Hanna M, Haugen DF, Juhl G, King S, Klepstad P, Laugsand EA, Maltoni M, Mercadante S, Nabal M, Pigni A, Radbruch L, Reid C, Sjogren P, Stone PC, Tassinari D, Zeppetella G; European Palliative Care Research Collaborative (EPCRC); European Association for Palliative Care (EAPC). Use of opioid analgesics in the treatment of cancer pain: evidence-based recommendations from the EAPC. Lancet Oncol. 2012 Feb;13(2):e58-68. doi: 10.1016/S1470-2045(12)70040-2. PMID 22300860
- [Background] Ahmedzai SH, Leppert W, Janecki M, Pakosz A, Lomax M, Duerr H, Hopp M. Long-term safety and efficacy of oxycodone/naloxone prolonged-release tablets in patients with moderate-to-severe chronic cancer pain. Support Care Cancer. 2015 Mar;23(3):823-30. doi: 10.1007/s00520-014-2435-5. Epub 2014 Sep 14. PMID 25218610
- [Background] Panchal SJ, Muller-Schwefe P, Wurzelmann JI. Opioid-induced bowel dysfunction: prevalence, pathophysiology and burden. Int J Clin Pract. 2007 Jul;61(7):1181-7. doi: 10.1111/j.1742-1241.2007.01415.x. Epub 2007 May 4. PMID 17488292
- [Background] Mueller-Lissner S. Fixed combination of oxycodone with naloxone: a new way to prevent and treat opioid-induced constipation. Adv Ther. 2010 Sep;27(9):581-90. doi: 10.1007/s12325-010-0057-y. Epub 2010 Aug 11. PMID 20714946
- [Background] Mancini I, Bruera E. Constipation in advanced cancer patients. Support Care Cancer. 1998 Jul;6(4):356-64. doi: 10.1007/s005200050177. PMID 9695203
- [Background] Kalso E. Oxycodone. J Pain Symptom Manage. 2005 May;29(5 Suppl):S47-56. doi: 10.1016/j.jpainsymman.2005.01.010. PMID 15907646
- [Background] Leppert W. Role of oxycodone and oxycodone/naloxone in cancer pain management. Pharmacol Rep. 2010 Jul-Aug;62(4):578-91. doi: 10.1016/s1734-1140(10)70316-9. PMID 20884999
- [Background] Stessel B, Theunissen M, Fiddelers AA, Joosten EA, Kessels AG, Gramke HF, Marcus MA. Controlled-release oxycodone versus naproxen at home after ambulatory surgery: a randomized controlled trial. Curr Ther Res Clin Exp. 2014 Nov 28;76:120-5. doi: 10.1016/j.curtheres.2014.10.001. eCollection 2014 Dec. PMID 25516773
- [Background] Salzman RT, Roberts MS, Wild J, Fabian C, Reder RF, Goldenheim PD. Can a controlled-release oral dose form of oxycodone be used as readily as an immediate-release form for the purpose of titrating to stable pain control? J Pain Symptom Manage. 1999 Oct;18(4):271-9. doi: 10.1016/s0885-3924(99)00079-2. PMID 10534967